CLINICAL TRIAL: NCT06777719
Title: Eight-Treg Study: a Phase I Dose Escalation Trial of Adoptive Immunotherapy With Autologous ex Vivo Expanded Regulatory CD8+ T Cells in Living Donor Kidney Transplant Recipients
Brief Title: Eight-Treg Study:Trial of Adoptive Immunotherapy With Autologous ex Vivo Expanded Regulatory CD8+ T Cells in Living Donor Kidney Transplant Recipients
Acronym: Eight-Treg
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: CR2TI, INSERM, UMR1064 (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC24_0033; 2024-513771-40-01 (EU CTIS Number)
Record Dates: First submitted 2024-12-23; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplantation; living donor kidney; immunotherapy; CD8+ T cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eight -Treg infusion Arm (Experimental): The experimental drug "Eight Treg"is given to patients with a peripheral IV infusion the day before the graft in addition to the maintenance protocol combining corticosteroids, tacrolimus and MPA which are classically pre-scribed in kidney graft patients from a living donor at the Nantes CHU.
  Interventions: Drug: Eight Treg

INTERVENTIONS:
Drug: Eight Treg — The experimental drug "Eight Treg" is given to patients with a peripheral IV infusion the day before the graft (cf section "5.1.5. "Infusion of the experimental drug" of this protocol) in addition to the maintenance protocol combining corticosteroids, tacrolimus and MPA which are classically pre-scribed in kidney graft patients from a living donor at the Nantes CHU.

SUMMARY:
The only curative treatment for end-stage renal disease is through kidney transplantation. Solid organ transplants success had been made possible by the development of Immunosuppressive (IS) drugs. However, the long-term survival of transplants is still shortened by the chronic dysfunction of the graft which is not prevented by current IS regimens. Moreover, these IS drugs increase the risk of opportunistic infections and malignancies, and have many non-immune side-effects that hamper their tolerability.

New research strategies are, therefore, developed with the aim of reducing the dependence on conventional pharmacological IS drugs. Regulatory cell therapy is one of these strategies. It consists of expanding specific populations of immune regulatory cells ex vivo into cell-based drugs that can then be infused into transplant recipients, with the goal of inducing graft tolerance.

This is the framework of this clinical trial. The experimental drug "Eight Treg" being evaluated in this study is an autologous cell therapy product containing CD8+ regulatory T lymphocytes (Tregs) expanded ex vivo during 21 days of cell culture. Team 2 of the Center for Research in Transplantation and Translational Immunology (CR2TI), Nantes University, INSERM, Mixed Research Unit (UMR) 1064, responsible for developing the manufacturing process of the experimental drug "Eight Treg", has demonstrated the feasibility of the expansion of CD8+ Tregs ex vivo and their ability to prevent skin graft rejection and inhibit Graft Versus Host Disease (GVHD) in NOD-Scid-IL-2γ-/- mouse models (NSG)14.

Based on the preclinical experience of CR2TI team 2, which has been working on basic and translational aspects of CD8+ Tregs for 15 years, the present phase I clinical trial aims to assess the safety of increasing doses of the experimental drug "Eight Treg" in 9 recipients of renal transplantation from a living donor. The possibility of manufacturing the experimental drug "Eight Treg" at the required doses, in accordance with the Good Manufacturing Process (GMP), has been assessed in validation runs as specified at the end of the "justification of the study" part of this protocol. This clinical trial will be the first administration of expanded CD8+ Tregs into humans, and it follows previous studies which evaluated the safety of other regulatory cell therapy products, containing expanded CD4+ Tregs and other regulatory cells (autologous tolerogenic dendritic cells performed by Nantes CHU laboratory and clinical services, for example), injected into patients in different contexts (renal transplantation, liver transplantation, GVHD, type 1 diabetes, etc) without causing any significant adverse effect. This study will pave the way for future, broader research on the use of CD8+ Tregs as a possible anti-rejection and tolerance inducer "drug" in transplantation.

ELIGIBILITY:
for kidney transplant recipient: pre-Inclusion Criteria:

1. Man or woman with chronic renal failure requiring kidney transplantation and approved to receive a primary kidney allograft from a living donor.
2. Weight between 50 and 100 kg.
3. Up-to-date vaccination against SARS Cov2 depending on the health situation and the rules in force with last recall done at least 6 to 1 month prior to visit 1.
4. Negative microlymphocytotoxicity (LCT) and flow cytometry crossmatches regardless of HLA compatibility
5. Signed and dated written informed consent *.
6. Aged at least of 18 years the day the consent is signed.
7. Able to commence the IS regimen at the protocol-specified time point.
8. As a precautionary measure, women of childbearing age should use an effective method of birth control, and male participants should use contraception to avoid partner pregnancy for the duration of the trial.
9. Affiliated or beneficiary of a social security scheme.
10. Speaking and understanding French.

Inclusion Criteria:

1. WOCBP must have a negative serum pregnancy test.
2. Respects the following conditions:

   * Condition 1: number of CD8+ Tregs / ml of blood > 2.096x106 CD8+ Tregs / weight
   * Condition 2 (depending on the dose level considered):

     * Dose 1: number of CD8+ Tregs / ml of blood > 1.15x104 CD8+ Tregs + 3.18x103 CD8+ Tregs / weight
     * Dose 2: number of CD8+ Tregs / ml of blood > 4.6x104 CD8+ Tregs + 3.18x103 CD8+ Tregs / weight
     * Dose 3: number of CD8+ Tregs / ml of blood > 9.22x104 CD8+ Tregs + 3.18x103 CD8+ Tregs / weight

Pre-Exclusion Criteria:

1. Patient has previously received any tissue or organ transplant other than the planned kidney graft.
2. Genetically identical to the prospective organ donor at the HLA loci.
3. Known contraindication to the protocol-specified treatments / medications or components used in the manufacture of the experimental drug.
4. Presence of donor-specific antibodies (DSA) detected prior transplantation determined by Luminex within 3 months or presence of cytotoxic DSA determined by cell-based CDC assay.
5. Previous treatment with any desensitisation procedure (with or without IVIg).
6. Concomitant malignancy or history of malignancy within 5 years prior to planned study entry (excluding successfully-treated non-metastatic basal / squamous cell carcinoma of the skin).
7. ABO incompatibility
8. Evidence of significant local or systemic infection on visit 1.
9. Malignant or pre-malignant haematological conditions.
10. Ongoing treatment with systemic IS drugs at visit 1 (except corticoids < 10 mg).
11. Any vaccine (or vaccine recall) dated within 3 months on visit 1 except the SARS Cov2*.
12. Participation in another clinical trial during the study or within 28 days prior to the planned study entry and / or exposure to an investigational product during the study or within 28 days prior to the planned study entry (date of signature of the consent collection form).
13. Women who are pregnant (or planning to be during the course of the study) or breastfeeding or women with a positive pregnancy test on enrolment (visit 1, screening failure).
14. Psychological, familial, sociological or geographical factors that potentially hampering compliance with the study protocol and follow-up visit schedule.
15. Any form of drug abuse, psychiatric disorder, or other condition that, in the opinion of the investigator, may invalidate communication with the investigator and/or designated study personnel.
16. Any pro-coagulant disposition, as evidences by a past history of thromboembolic disease or abnormal laboratory coagulation parameters which, in the judgement of the investigator, would place the subject at undue risk.
17. Any condition resulting in a substantial reduction in the volume of the pulmonary vasculature or an increase in the pulmonary vascular resistance. Any disease or disease process leading to substantially elevated pulmonary arterial pressure (as evidences by electrocardiography, echocardiography, radiology or cardiac catheterization) or right heart hypertrophy or dysfunction.
18. Known atrial or ventricular septal defects posing a risk of paradoxical embolism of infused cells or cell aggregates.
19. Patients unable to freely give their informed consent (e.g. patients under guardianship, curatorship, protection of justice).
20. Patients deprived of their liberty.

Exclusion Criteria:

1. Human Immunodeficiency Virus (HIV)-positive, Epstein-Barr Virus (EBV)-negative (if donor is EBV positive), HTLV positive, syphilis-positive serology or suffer from chronic viral hepatitis.
2. Significant liver disease, defined as persistently elevated Aspartate Transaminase (AST) and / or Alanine Transaminase (ALT) levels > 2 x upper limit of normal range.

Donor:

Pre-Inclusion Criteria:

1. Willing and able to provide a blood and an urine sample for the immune monitoring.
2. Willing to provide personal and medical/biological data for the trial analysis.
3. Signed and dated written informed consent *.
4. Aged at least of 18 years the day the consent is signed.
5. Affiliated or beneficiary of a social security scheme.
6. Speaking and understanding French.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 up to 3 months post-graft | 3 months
Occurrence of a dose-limiting toxicity, defined as the occurrence of an AE of grade 3 or higher (with exceptions: see specific section) up to visit 10, at 3 months post-transplantation. | 3 months

SECONDARY OUTCOMES:
Number of participants with the (absence or low) occurrence of a dose limiting toxicity at 6 and 12 months post-graft | 12 months
Number of participants with the (no or low stage of) graft inflammation at 3-months post-graft | 3 months
Number of participants with the (lower) total immunosuppressive burden at one post-transplant year | 12 months
Number of participants with the (lower) incidence, duration and severity of infections during the first year post-graft compared to historical data from previously reported studies | 12 months
Biological evaluation of the impact of CD8+ Treg cell therapy on immune response by real time follow-up of blood cell count by flow cytometry (FC) to evaluate and characterize cellular and humoral immune responses towards the graft | 12 months
Comparison of Tregs profile and clones emerging in the "Eight-Treg" group by scRNAseq and VDJseq compared to reference group | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided